CLINICAL TRIAL: NCT03489811
Title: The Effect of Aroma on Anxiety Among Children With Autism.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic introduced confounding factors that would bias the study data. Study rescheduled for future dates post-pandemic.
Sponsor: Nutraceuticals Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17-2100
Record Dates: First submitted 2018-03-30; First posted 2018-04-06 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Anxiety; Autism Spectrum Disorder
Keywords: Essential Oils; Aromatherapy; Anxiety; Autism Spectrum Disorder
MeSH Terms: conditions — Anxiety Disorders; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Essential Oil Blend (Experimental): Participants in this arm receive the test essential oil inhaler to administer during the 4-week intervention.
  Interventions: Other: Test Essential Oil Blend
- Active Essential Oil Blend (Active Comparator): Participants in this arm receive an active essential oil inhaler to administer during the 4-week intervention.
  Interventions: Other: Active Essential Oil Blend
- Control (Placebo Comparator): Participants in this arm receive a control inhaler to administer during the 4-week intervention.
  Interventions: Other: Control Blend

INTERVENTIONS:
Other: Test Essential Oil Blend — The test essential oil blend consists of plant derived oils which have been distilled from crude plant matter and analyzed in a laboratory to identify chemical composition.
  Arms: Test Essential Oil Blend
Other: Active Essential Oil Blend — The active essential oil blend consists of plant derived oils which have been distilled from crude plant matter and analyzed in a laboratory to identify chemical composition.
  Arms: Active Essential Oil Blend
Other: Control Blend — The control blend consists of inert vegetable oils which are produced from plant matter.
  Arms: Control

SUMMARY:
This study evaluates the effects of essential oils on anxiety scores among children who have an autism spectrum disorder. One third of the children will receive a control blend of oils, one third of the children will receive a test blend of oils, and the other third will receive a second test blend of oils.

DETAILED DESCRIPTION:
Essential oils have been found in studies to reduce both stress and anxiety as measured by an anxiety inventory, but studies have not tested these effects among children who have an autism spectrum disorder.

The essential oils used in this study are administered each morning for a total period of four weeks, with an optional second exposure on an as-needed basis during the final two of the four weeks of the study. The oils are administered during this time to evaluate both the preventive effects and the treatment effects of the essential oils.

Anxiety is measured on an anxiety inventory, which is completed by the parent of the participant at the end of each week during the study. Parents complete this data online, allowing them to participate from anywhere in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* age: 6-11 years old at enrollment
* diagnosed with an autism spectrum disorder

Exclusion Criteria:

* mast cell activation syndrome
* history of adverse response to essential oil inhalation

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
39-Question Spence Children's Anxiety Scale (SCAS) | baseline and day 35
  The Spence Children's Anxiety Scale collects parent-reported signs and symptoms of anxiety at baseline and again at the end of each week of the intervention. Each item is scored as (0) never, (1) sometimes (2) often, or (3)always. The total score ranges from 0-114, with higher scores indicating higher levels of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Franklin Institute of Wellness, Franklin, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared.